CLINICAL TRIAL: NCT07080177
Title: Assessment of Hard and Soft Tissue Changes Following Xenogeneic Collagen Membrane Versus Free Gingival Graft Simultaneous With Delayed Dental Implant Placement: Randomized Controlled Clinical Trial
Brief Title: Assessment of Hard and Soft Tissue Changes Following XCM Versus FGG Simultaneous With Delayed Dental Implant Placement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: MTI University (Other)
Responsible Party: Principal Investigator, Parryhan Mohamed Abdelsamie, Lecturer of periodontology, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTI
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Missing Teeth
Keywords: xenogeneic collagen membrane; free gingival graft; xenogeneic collagen matrices; simultaneous implant placement
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xenogeneic collagen matrix simultaneous with delayed implant placement (Experimental): Tissue punch technique implants will be placed. XCM grafts (of bovine origin) will be trimmed to the required dimensions and will be fixed to the periosteum and sutured to the buccal peri-implant mucosa
  Interventions: Procedure: Xenogeneic collagen matrix simultaneous with delayed implant placement
- Free gingival graft simultaneous with delayed implant placement (Active Comparator): Tissue punch technique implants will be placed. A FGG will be harvested from the palate then the outlined graft will be placed and sutured to the recipient bed of the buccal peri-implant mucosa
  Interventions: Procedure: Free gingival graft simultaneous with delayed implant placement

INTERVENTIONS:
Procedure: Free gingival graft simultaneous with delayed implant placement — XCM grafts (of bovine origin)
  Arms: Free gingival graft simultaneous with delayed implant placement
Procedure: Xenogeneic collagen matrix simultaneous with delayed implant placement — A FGG will be harvested from the palate between first premolar and first molar
  Arms: Xenogeneic collagen matrix simultaneous with delayed implant placement

SUMMARY:
Teeth loss are usually associated with alterations of extraction sockets result in obviously absorbed alveolar ridges and are often accompanied with soft tissue atrophy such as narrow keratinized tissue and a shallow vestibule.

Lack of peri-implant keratinized tissue is a potential risk to peri-implant diseases. Although the role of width of KM in maintaining peri-implant health is a controversial topic, the majority of high-level evidence has suggested that a minimum KM width (KMW) of 2 mm around the dental implants is critical to maintain peri-implant health and the long-term survival of dental implants.

DETAILED DESCRIPTION:
This study will be carried out on patients attending outpatient clinic of Oral maxillofacial surgery and Periodontology Departments, Faculty of Dentistry. Modern University for Technology and Information, Cairo, Egypt.

P: Healthy patients with posterior missing teeth with deficient keratinized tissue to receive delayed dental implant placement I: Xenogeneic collagen membrane (XCM) simultaneous with delayed implant placement C: Free gingival graft (FGG) simultaneous with delayed implant placement O: Keratinized tissue width (KMW), graft shrinkage (GS), marginal bone loss (MBL) T- One year S- Randomized controlled clinical trial.

Eligible patients will be divided into equal proportions between control group and test group.

The control group "Group 1" will receive FGG simultaneous with implant placement The test group "Group 2" will receive XCM simultaneous with implant placement

ELIGIBILITY:
Inclusion Criteria:

1. Adults above the age of 18 years.
2. Presence of 2mm or less of keratinized tissue width
3. Sufficient alveolar ridge width minimum of 6 mm
4. Patients with good oral hygiene as evidenced by plaque index (PI)<1 and showing cooperation or compliance with treatment.

Exclusion Criteria:

1. Patients diagnosed with periodontal diseases (Caton et al., 2018).
2. Acute active infection at implant sites
3. Patients with medical conditions that would compromise the surgical procedures; uncontrolled diabetes mellitus, taking intravenous bisphosphonates for treatment of osteoporosis and radiotherapy
4. Patients with parafunctional habits.
5. Smokers (≥10 cigarettes per day),

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Keratinized tissue width | One year
  mm
graft shrinkage | One year
  precentage
marginal bone loss | One year
  mm

CONTACTS AND LOCATIONS:
Overall Officials: Parryhan M Abdelsamie, PhD, Principal Investigator — MTI University; Maged M Seleet, PhD, Principal Investigator — MTI University
Locations (1):
- MTI University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No